CLINICAL TRIAL: NCT02762916
Title: Randomized Trial of CONTECI Program: Pilot Study
Brief Title: CONTECI Program: A New Way to Control Peripheral Arterial Disease Using New Technologies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Consorci Sanitari del Maresme (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 18/14
Record Dates: First submitted 2016-04-28; First posted 2016-05-05 (Estimated); Last update posted 2016-05-05 (Estimated); Status verified 2016-05

CONDITIONS: Peripheral Arterial Disease; Personal Satisfaction; Telemedicine
MeSH Terms: conditions — Peripheral Arterial Disease; Personal Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1- Telemedicine arm (Experimental): The intervention arm (IA), telehealth control, were followed up by himself helped by CONTECI program. They have to use every three months and if somethings was wrong the patient have to send mail to the doctor.
  The intervention consisted to use the CONTECI program (included test) for the following of the patients.
  Interventions: Other: Selfmanage with the help of telemedicine program
- 2- Control arm (No Intervention): The Control Arm (CA) were followed up as usual every 6 months in outpatient vascular visits in the clinical hospital. If some patient have a complications or and emergency they have to do usual protocol, go to primary care or emergency.

INTERVENTIONS:
Other: Selfmanage with the help of telemedicine program — The intervention group patients were not followed by the usual protocol, but it used the program CONTECI (and test different directions) to guide the patient monitoring.
  Both groups used antiplatelets and statines as usual protocol (these were not the interventions) We did not use drugs or device for the intervention, only a Telemedicine programme
  Arms: 1- Telemedicine arm

SUMMARY:
The current increase in chronic diseases calls for changes to the health system. It is necessary to promote expert patient in chronic disease. The expansion of new technologies gives us new tools to face new challenges, providing efficiency, expertise and autonomy. The characteristics of peripheral arterial disease make possible to promote expert patient and the self-management. In order to bring these concepts together the telemedicine program was created to promote expert patient for increasing the quality of life and satisfaction of patients and improving the efficiency of the health system.

Methods: Randomized clinical trial on patients with peripheral arterial disease in intermittent claudication grade. They were randomized into two groups: intervention arm (IA) using CONTECI program for self-managing and control arm (CA), followed as usual vascular visits.

ELIGIBILITY:
Inclusion Criteria:

* Patient with confirmed PAD
* Over 18 years old
* Informed Consent
* Internet Access (patient or family)
* Spanish or Catalan fluidity

Exclusion Criteria:

* Cognitive impairment
* Previous patency arterial surgery
* Sever chronic obstructive pulmonary disease (GOLD III/ IV)
* Patients with decreased survival of 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2014-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
satisfaction. Analogical scale 0-100. To compare the satisfaction in the new model control and the model before | 12 months

SECONDARY OUTCOMES:
Clinical features. Pateint who turned to grade 3 or 4 of Le Fontaine classification, number of surgeries. | 6 and 12 months
  PAD grade 3 and 4, surgeries
Health resources consumption: rate of Emergency visits, scheduled visits, extra visits, Mail per participant | 6 and 12 months
Quality of life. EuroQol5D were used. Change from baseline Quality of line at 12 months. | 12 months

IPD SHARING:
Plan to Share IPD: No